CLINICAL TRIAL: NCT03122600
Title: Ankle Brachial Index (ABI) Versus Conventional Cardiac Risk Indices To Predict Cardiac Affection In High Risk Patients Under General Anesthesia
Brief Title: Ankle Brachial Index Versus Conventional Cardiac Risk Indices
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Sayed Abd El Aal, assistant lecturer, Assiut University
Other Study IDs: IRB0000
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vascular surgery group: Elderly patients undergoing vascular surgery in the lower half of the body

SUMMARY:
the applicability of ankle brachial index (ABI) and B-type natriuretic peptide (BNP) measurement as cardiovascular risk prediction models during hospital stay in elderly patients undergoing vascular surgery.

DETAILED DESCRIPTION:
A major public health challenge is therefore to accurately identify, in an apparently healthy population, those who are at high risk and to target prevention at these individuals. Although primary prevention measures, including aspirin, have been suggested for all individuals with an estimated intermediate to high cardiovascular risk of 2% per year, the best method of identifying such individuals has not been established. In addition, models based on conventional risk factors have been shown to have limited predictability and several restrictions. They were not designed for people with preexisting cardiovascular disease (CVD), and when risk factors are at extreme levels, the equations may underestimate or overestimate risk. In this regard, interest is increasing in the use of noninvasive markers that allow the identification of sub-clinical atherosclerosis, including the ankle brachial index (ABI), ratio of ankle to arm systolic blood pressure). Although quick and easy to perform with a high patient acceptability, the ABI was originally used to identify lower-limb atherosclerosis. However, it has subsequently been shown to be an accurate and reliable marker of generalized atherosclerosis. Cohort studies between 5 and 10 years of follow-up have shown that people with a low ABI have an increased risk of both cardiovascular morbidity and mortality. They have previously reported that the 5-year incidence of total cardiovascular events in subjects with an ABI ˂ 0.9 was almost twice that in subjects with an ABI ˃ 0.9 Furthermore, examination of positive predictive values showed that a low ABI was better at predicting risk of future cardiovascular and cerebrovascular events than conventional risk factors alone.

B-type natriuretic peptide (BNP) is a cardiac neuro-hormone secreted from membrane granules in the cardiac ventricles as a response to ventricular volume expansion and pressure overload. The natriuretic peptide system allows the heart to participate in the regulation of vascular tone and extracellular volume status. The natriuretic peptide system and the renin angiotensin system counteract each other in arterial pressure regulation. Levels of atrial natriuretic peptide (ANP) and B-type natriuretic peptide (BNP) are elevated in cardiac disease states associated with increased ventricular stretch. The main circulating and storage form of BNP is 32 amino acid peptide with a ring structure. Physiological actions of BNP are mediated through a guanylate cyclase-linked receptor, natriuretic peptide receptor A (NPR-A). BNP produces arterial and venous vasodilatation. Clearance of BNP is promoted by a natriuretic peptide receptor C (NPR-C) which removes it from the circulation and BNP is also degraded through enzymatic cleavage by neutral endopeptidase. BNP levels are reflective of left ventricular diastolic filling pressures and thus correlate with pulmonary capillary wedge pressure.

BNP levels have been shown to be elevated in patients with symptomatic left ventricular dysfunction and correlate with New York Heart Association (NYHA) classification and prognosis.

Based on the available information a BNP < 100 pg/ml, allows clinicians to exclude heart failure as a cause of the patients' symptoms or physical exam signs in most circumstances BNP levels have been shown to predict long term mortality in patients with heart failure, independent of other established prognostic variable

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years or older
* American Society of Anesthesiologists (ASA) III or IV
* Operation in the lower half of the body

Exclusion Criteria:

* Patient refusal
* Patient with acute cardiac condition (MI, recent MI ,sever valve lesion or heart failure)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients, undergoing vascular surgery in the lower half of the body under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
myocardial ischemia | up to 7 days postoperative
  incidence of myocardial ischemia after operation

SECONDARY OUTCOMES:
myocardial infarction | up to 7 days postoperative
  incidence of myocardial infarction after operation
mortality | up to 7 days postoperative
  incidence of mortality related to cardiac problems

CONTACTS AND LOCATIONS:
Overall Officials: Esam Abd Allah, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided